CLINICAL TRIAL: NCT02302560
Title: Identification of the Sleep Architecture in Patients With Hip Surgery (TepSo)
Status: Withdrawn | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Univ.-Prof. Dr. C. Spies, Charite University, Berlin, Germany
Other Study IDs: TepSo
Record Dates: First submitted 2014-11-07; First posted 2014-11-27 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Sleep Architecture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with elective hip surgery: Patients with elective hip surgery (implementation or replacement of hip joint endoprotheses).

SUMMARY:
The purpose of this prospective observational study is to investigate the changes in sleep architecture after a hip surgery and its potential association with postoperative delirium and postoperative cognitive dysfunctions respectively.

DETAILED DESCRIPTION:
Sleep research has confirmed the association of sleep (REM sleep and slow-wave sleep) with memory and cognitive function in general. There are changes in the quantity of REM sleep after certain forms of anesthesia, especially with barbiturate, as shown in mouse model. This study is designed to be the first explorative clinical studyl to measure changes in sleep architecture in surgical patients undergoing different types of anesthesia (general anesthesia and spinal anesthesia) and its potential associations with the development of postoperative delirium and postoperative cognitive dysfunction. Additionally, parameters will be collected, that from recent research are suspected to be reliable markers for systemic inflammation that might account for delirium and cognitive dysfunction after surgical interventions.

Patients were stratified into two groups: age (≤ 65 years; > 65 years) and benzodiazepine premedication (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age 50 years and above
* Intervention for hip joint endoprosthesis or replacement of endoprosthesis at the Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum, Charité - University Medicine Berlin

Exclusion Criteria:

* Lacking willingness to save and hand out data within the study
* Missing informed consent of the patient
* Participation in other prospective interventional study 10 days before study inclusion and during the study period
* Patients with diagnosed and treated sleep disorders
* Patients with psychiatric diseases
* Patients with injuries or operations of the enteral tract and the esophagus respectively in the last four weeks before the hip surgery
* Allergies to any substance of the electrode fixing material
* Dermatoses in the area of the electrodes to be fixed

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with elective hip surgery (implementation or replacement of hip joint endoprothesis)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Changes in prevalence of rapid eye movement sleep | Up to 36 hours
  Changes in prevalence of rapid eye movement (REM) sleep in the preoperative night compared to the night following the first postoperative day, including potentially compensatory sleep during daytime after surgery.
  Sleep architecture will be measured with the Somnoscreen device for mobile polysomnography for a total time duration of 36 h (beginning in the preoperative evening, to be finished the morning of the second postoperative day).

SECONDARY OUTCOMES:
Insomnia Severity Index | Up to 90 days after the operation
  The ISI will be assessed by self-assessment questionnaire
Malnutrition | Up to 90 days after the operation
  Malnutrition Screening Tools
Epsworth Sleepiness Scale | Up to 90 days after the operation
  The ESS will be assessed by self-assessment questionnaire
Postoperative Cognitive Dysfunction | Up to 90 days after the operation
  Postoperative Cognitive Dysfunction will be measured at hospital discharge and at the 90th postoperative day.
Depth of anesthesia | At time of surgery
  Depth of anesthesia will be measured by processive Electroencephalography and Electromyography (EEG/EMG) -Data (SedLine®)
Opioid requirements | Participants will be followed up for hospital stay an expected average of 7 days
  Postoperative pain will be measured by Numeric Rating Scale - Visualized (NRS-V), the Faces Pain Scale - Revised (FPS-R), the Behavioral Pain Scale (BPS) or the Behavioral Pain Scale for Non-Intubated (BPS-NI)
Length of hospital stay | Participants will be followed up for hospital stay an expected average of 7 days
Pain | Participants will be followed up for hospital stay an expected average of 7 days
  Postoperative pain will be measured by Numeric Rating Scale - Visualized (NRS-V), the Faces Pain Scale - Revised (FPS-R), the Behavioral Pain Scale (BPS) or the Behavioral Pain Scale for Non-Intubated (BPS-NI)
N-Methyl-D-aspartate (NMDA)-receptor autologous antibodies | Up to 90 days after the operation
  Identification of NMDA-receptor autologous antibodies in blood serum and cerebrospinal fluid; the requested blood samples will be collected on the operation day, on the last day of hospitalisation and after 90 days. The requested liquor samples will be collected on the operation day (only in patients with spinal anesthesia).
Inflammation parameters | Participants will be followed up for hospital stay an expected average of 7 days
  Assessment of inflammation parameters by means of extended differential blood count (Sysmex) ; the requested blood samples will be collected on the preoperative day, on the day of the intervention, on the following day and on the last day of the hospitalisation
Hemodynamic parameters | At time of surgery
  Hemodynamic variables are assessed by the anesthesia monitor and esophageal Doppler Monitor
Changes in prevalence of rapid eye movement sleep | Up to 24 hours
  REM-Sleep at operation day/night in comparison to preoperative night. Sleep architecture will be measured with the Somnoscreen device for mobile polysomnography for a total time duration of 24 h.
Changes in prevalence of slow-wave sleep (Stadium 3 of non rapid eye movement-sleep) | Up to 24 hours
  Slow wave sleep at operation day/night in comparison to preoperative night. Sleep architecture will be measured with the Somnoscreen device for mobile polysomnography for a total time duration of 24 h.
Changes in prevalence of slow-wave sleep (Stadium 3 of non rapid eye movement-sleep) | Up to 36 hours
  Changes in prevalence of slow-wave sleep in the preoperative night compared to the night following the first postoperative day, including potentially compensatory sleep during daytime after surgery.
  Sleep architecture will be measured with the Somnoscreen device for mobile polysomnography for a total time duration of 36 h (beginning in the preoperative evening, to be finished the morning of the second postoperative day).
Postoperative complications | Participants will be followed up for hospital stay an expected average of 7 days
  Including Severity of Delirium
Transfusion requirements | Participants will be followed up for hospital stay an expected average of 7 days
Catecholamine administration intra- und postoperative | Participants will be followed up for hospital stay an expected average of 7 days
Severity of postoperative Delirium | Up to 36 hours
  Delirium screening will be conducted preoperatively, one hour postoperative, the evening of operation day, and the following morning with the scoring devices of confusion assessment method (CAM), by confusion assessment method in the intensive care unit (CAM-ICU) or by Nursing Delirium Screening Scale (Nu-DESC)

OTHER OUTCOMES:
Tissue Inhibitor of Metalloproteinases | At time of spinal anesthesia
  Metalloproteinases (MMP-2 und MMP-9) from liquor samples (only in patients with spinal anesthesia).
Metalloproteinases | At time of spinal anesthesia
  Metalloproteinases (MMP-2 und MMP-9) from liquor samples (only in patients with spinal anesthesia).
ASA (physical status classification system) status | At the beginning of the investigation
Benzodiazepine premedication | At the beginning of the investigation

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Berlin, Berlin, Germany